CLINICAL TRIAL: NCT05550545
Title: ResQ Family: Impact of Respiratory Syncytial Virus (RSV) Hospitalisation on Quality of Life of Families - A Multi-Country Study
Brief Title: Infant RSV Infections and Health-related Quality of Life of Families
Acronym: ResQFamily
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Global Foundation for the Care of Newborn Infants (Other)
Collaborators: Respiratory Syncytial Virus Foundation (ReSViNET) (Unknown); European Society for Paediatric Research (ESPR) (Unknown); Union of European Neonatal and Perinatal Societies (UENPS) (Unknown)
Responsible Party: Principal Investigator, Johanna Kostenzer, Head of Scientific Affairs, Global Foundation for the Care of Newborn Infants
Other Study IDs: 2022-3307
Record Dates: First submitted 2022-09-12; First posted 2022-09-22 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: RSV Infection; Quality of Life; Infant ALL; Caregiver Burden; Family
Keywords: RSV; Respiratory syncytial virus; quality of life; health literacy; infants; children; caregiver burden
MeSH Terms: conditions — Respiratory Syncytial Virus Infections; Caregiver Burden | interventions — Cohort Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parents/caregivers of RSV-infected infants
  Interventions: Other: cohort study

INTERVENTIONS:
Other: cohort study — Please note that this is an observational study; not applicable

SUMMARY:
Until today, there is only little information available on how severe RSV infection leading to hospitalisation of the infant impacts the quality of life of affected families. For the ResQ Family project, an online questionnaire will be used to survey parents or caregivers of children up to 24 months currently or recently hospitalised (length of hospital stay of at least 12 hours and hospital admission no longer than 4 weeks ago) due to RSV infection.

The aim of the ResQ Family project is to find out how infant RSV hospitalisation impacts the quality of life of affected children and their families. The goal is further to provide scientific evidence on the burden of RSV and raise awareness among all relevant stakeholders including healthcare professionals and patient representatives, decision-makers and the general public. The project will run until June 2024. Data collection will take place during the RSV season from fall 2022 to spring 2023 in four European countries: France, Germany, Italy, and Sweden.

DETAILED DESCRIPTION:
Respiratory Syncytial Virus (RSV) is a very contagious virus and the most common cause of lower respiratory tract infections such as bronchiolitis and pneumonia in infants. By the age of two years, nearly all infants will be infected with RSV at least once. Globally, it is a leading cause of hospitalisations among young infants with approximately 33 million cases of acute lower respiratory infections causing more than three million hospitalisations each year in children younger than 5 years. While most RSV cases are mild, one can't predict which infants could get seriously ill and end up in hospital. This is because the course of the disease is unpredictable.

When the RSV infection of the child is severe and associated with hospitalisation, it may lead to intensive care unit admissions with use of supportive care such as mechanical ventilation. It may further result in long-term complications such as recurrent wheezing, reduced pulmonary function and asthma. Moreover, RSV-related hospitalisations can be associated with a significant burden on the entire family, causing considerable stress and increased loss of work productivity. Currently, there is a lack of adequate information on how severe RSV infection leading to hospitalisation of infants (< 2 years) impacts the quality of life of affected families.

To close this knowledge gap, the ResQ Family research project was initiated: ResQ Family: Impact of Respiratory Syncytial Virus (RSV) hospitalisation on Quality of life of Families - a multi-country study. The project runs from December 2021 until June 2024 and covers four European countries: France, Germany, Italy and Sweden. Data will be collected between autumn 2022 and spring 2023, corresponding to a typical RSV season duration in temperate countries in the northern hemisphere.

The aim of the ResQ Family study is to find out how infant RSV hospitalisation impacts the quality of life of affected children and their families. The goal is further to provide scientific evidence on the burden of RSV and raise awareness among all relevant stakeholders including healthcare professionals and patient representatives, decision-makers and the general public.

An online questionnaire will be used to ask parents and caregivers of children experiencing (or having recently experienced) hospitalisation due to RSV infection to share their experiences and a follow-up will take place after six weeks. The study focuses on children up to 24 months with a hospital stay due to RSV infection of at least 12 hours in total. The hospital admission should not be longer than 4 weeks ago.

Experienced researchers and health care professionals renowned in the field of RSV as well as parent/patient representatives support the project as part of an external scientific advisory board and a project expert group.

EFCNI received a research grant from Sanofi in support of this independent study.

ELIGIBILITY:
Inclusion Criteria:

* Parents or caregivers of children younger than 24 months of age with a hospitalisation for at least 12 hours due to RSV infection
* Living in Germany, Sweden, Italy or France
* The diagnosis can either be confirmed by a test such as ELISA/IFT/PCR from nasal secretion, sputum or throat swab or by a doctor based on specific symptoms typically during the RSV season
* They can be reached during or after hospitalisation, ideally right after the discharge from hospital but at least within four weeks after hospital admission

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Parents or caregivers of children younger than 24 months of age with a hospitalisation for at least 12 hours due to RSV infection in Germany, Sweden, Italy or France.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-09-29 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life of parents/caregivers and family functioning | Baseline (Day 0)
  The 36-item version of the Pediatric Quality of Life Inventory Family Impact Module (PedsQLTM FIM) was used to assess the quality of life of parents/caregiver when the child was infected and hospitalized for RSV. It composes of six scales measuring parent self-reported functioning: 1) Physical functioning (6 items), 2) Emotional functioning (5 items), 3) Social functioning (4 items), 4) Cognitive functioning (5 items), 5) Communication (3 items), 6) Worry (5 items), and in addition two scales measuring parent-reported family functioning: 7) Daily activities (3 items) and 8) Family relationships (5 items). Each of the items have five Likert response options: 0 = never a problem, 1 = almost never, 2 = sometimes, 3 = often, 4= almost always. Items are reverse-scored and linearly transformed to a 0-100 scale (0 = 100, 1 = 75, 2 = 50, 3 = 25, 4 = 0), so that higher scores indicate better functioning (less negative impact).
Health-related quality of life of parents/caregivers and family functioning | 6 weeks follow-up (Week 6)
  The 36-item version of the Pediatric Quality of Life Inventory Family Impact Module (PedsQLTM FIM) was used to assess the quality of life of parents/caregiver when the child was infected and hospitalized for RSV. It composes of six scales measuring parent self-reported functioning: 1) Physical functioning (6 items), 2) Emotional functioning (5 items), 3) Social functioning (4 items), 4) Cognitive functioning (5 items), 5) Communication (3 items), 6) Worry (5 items), and in addition two scales measuring parent-reported family functioning: 7) Daily activities (3 items) and 8) Family relationships (5 items). Each of the items have five Likert response options: 0 = never a problem, 1 = almost never, 2 = sometimes, 3 = often, 4= almost always. Items are reverse-scored and linearly transformed to a 0-100 scale (0 = 100, 1 = 75, 2 = 50, 3 = 25, 4 = 0), so that higher scores indicate better functioning (less negative impact).

SECONDARY OUTCOMES:
Socio-demographics | Baseline (Day 0)
  Parental self-report - self-designed questions: socio-demographics (parents/caregiver), risk factors (smoking, allergic diseases), place of living, birth weight (child, categories and in grams), RSV prophylaxis, breastfeeding, day-care attendance
Child's co-morbidities | Baseline (Day 0)
  Parental self-report - self-designed questions: pre-existing health-conditions before or apart from the current recent hospitalisation due to RSV
Child's symptoms during RSV infection and hospitalisation | Baseline (Day 0)
  Parental self-report - self-designed questions:
  RSV diagnose (child), duration of hospitalisation (in days), supportive care measure in hospital, feelings (parents) in relation to the hospitalisation of the child (categories), presence with the child receiving special/intensive care, duration of symptoms (up to 7 days and more), child's behaviour (categories), worry of parents/caregiver about symptoms (categories)
Child's symptoms after RSV infection and hospitalisation | 6 weeks follow-up (Week 6)
  Parental self-report - self-designed questions:
  Duration of symptoms (in days), child's behaviour, worry of parents/caregiver about symptoms (categories)
Other | Baseline (Day 0)
  Parental self-report - self-designed questions:
  Health literacy, support structures, loss of work productivity (in hours), subjective assessment of parental health status (categories: 1=very bad to 10 = excellent), overall impact of the entire RSV episode (open question)
Other | 6 weeks follow-up (Week 6)
  Parental self-report - self-designed questions:
  Loss of work productivity (in hours), subjective assessment of parental health status (categories: 1=very bad to 10 = excellent), overall impact of the entire RSV episode (open question)

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Kostenzer, PhD, Principal Investigator — Global Foundation for the Care of Newborn Infants
Locations (1):
- EFCNI, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Trautmannsberger I, Plagg B, Adamek I, Mader S, de Luca D, Esposito S, Silfverdal SA, Zimmermann LJI, Tischer C; ResQ Family study group. The Multifaceted Burden of Respiratory Syncytial Virus (RSV) Infections in Young Children on the Family: A European Study. Infect Dis Ther. 2024 Jul;13(7):1531-1573. doi: 10.1007/s40121-024-00989-0. Epub 2024 May 20. PMID 38767780